CLINICAL TRIAL: NCT05611177
Title: Predicting Mortality in Patients With the Acute Respiratory Distress Syndrome Using Machine Learning
Brief Title: Predicting ICU Mortality in ARDS Patients
Acronym: POSTCARDS
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Jesus Villar, principal investigator, Dr. Negrin University Hospital
Other Study IDs: 7/2021
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: outcome; mechanical ventilation; intensive care unit; machine learning
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Logistic Models

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Derivation cohort: It will contain 700 patients (70% of 1000 ARDS patients)
  Interventions: Other: machine learning analysis
- Validation cohort: It will contain 300 patients (30% of 1000 ARDS patients)
  Interventions: Other: machine learning analysis
- Confirmatory cohort: It will contain 303 patients (for external validation)
  Interventions: Other: machine learning analysis

INTERVENTIONS:
Other: machine learning analysis — We will use robust machine learning approaches, such as Random Forest, XGBoost or Neural Networks.
  Other Names: Logistic regression; cross-validation; are aunder the ROC curves

SUMMARY:
The investigators are planning to perform a secondary analysis of an academic dataset of 1,303 patients with moderate-to-severe acute respiratory distress syndrome (ARDS) included in several published cohorts (NCT00736892, NCT02288949, NCT02836444, NCT03145974), aimed to characterize the best early model to predict duration of mechanical ventilation and mortality in the intensive care unit (ICU) after ARDS diagnosis using machine learning approaches.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is a severe form of acute hypoxemic respiratory failure in Critical Care Units worldwide. Most ARDS patients requiere mechanical ventilation (MV). Few studies have investigated the prediction of MV duration and mortality of ARDS.

For model description, the investigators will extract data from the first two ICU days after diagnosis of moderate-to-severe ARDS from patients included in the de-identified database, which includes 1,303 mechanically ventilated patients enrolled in several observational cohorts in Spain, coordinated by the principal investigator (JV), and funded by the Instituto de Salud Carlos III (ISCIII). The investigators will follow the TRIPOD guidelines and machine learning tecniques will be implemented (Random Forest, XGBoost, Logistic regression analysis, and/or neural networks) for development of the prediction model, and the accuracy will be compared to those of existing scoring systems for assessing ICU severity (APACHE II, SOFA) and the PaO2/FiO2 ratio. For external validation, the investigators will use 303 patients enrolled in a contemporary observational study (NCT03145974). The investigators will evaluate the accuracy of prediction models by calculating the respective confusion matrices and several statistics such as sensitivity, specificity, positive predictive value, and negative predictive value for mortality and duration of MV. Investigators will select the best probabilistic model with a minimum number of clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Berlin criteria for moderate to severe ARDS

Exclusion Criteria:

* Postoperative patients ventilated <24h; brain death patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: De-identified dataset including 1,303 patients with moderate/severe ARDS admitted consecutively in a network of Spanish ICUs.
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
ICU mortality | up to 6 months
  mortality in the intensive care unit

SECONDARY OUTCOMES:
MV duration | from ARDS diagnosis to extubation
  Duration of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, PhD, Principal Investigator — Hospital Universitario D. Negrin
Locations (3):
- Spain (3):
  - Hospital Universitario Dr. Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Department of Anesthesia, Hospital Clinic, Barcelona
  - Hospital Universitario La Paz (ICU), Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villar J, Ambros A, Mosteiro F, Martinez D, Fernandez L, Ferrando C, Carriedo D, Soler JA, Parrilla D, Hernandez M, Andaluz-Ojeda D, Anon JM, Vidal A, Gonzalez-Higueras E, Martin-Rodriguez C, Diaz-Lamas AM, Blanco J, Belda J, Diaz-Dominguez FJ, Rico-Feijoo J, Martin-Delgado C, Romera MA, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. A Prognostic Enrichment Strategy for Selection of Patients With Acute Respiratory Distress Syndrome in Clinical Trials. Crit Care Med. 2019 Mar;47(3):377-385. doi: 10.1097/CCM.0000000000003624. PMID 30624279
- [Background] Huang B, Liang D, Zou R, Yu X, Dan G, Huang H, Liu H, Liu Y. Mortality prediction for patients with acute respiratory distress syndrome based on machine learning: a population-based study. Ann Transl Med. 2021 May;9(9):794. doi: 10.21037/atm-20-6624. PMID 34268407